CLINICAL TRIAL: NCT03989817
Title: The Effects of a Long-lasting Infusion of Vasoactive Intestinal Peptide (VIP) on Headache, Cranial Hemodynamic in Healthy Volunteers
Brief Title: The Effects of a Long-lasting Infusion of Vasoactive Intestinal Peptide (VIP) on Headache, Cranial Hemodynamic and Autonomic Symptoms in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, MD, PhD student, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: VIP H-18050862
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Headache Disorders
MeSH Terms: conditions — Headache Disorders | interventions — Vasoactive Intestinal Peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIP (Active Comparator): To investigate the role of VIP on cranial hemodynamic and headache in healthy volunteers.
  Interventions: Drug: Vasoactive Intestinal Peptide (VIP) and Saline
- Saline (Placebo Comparator): To investigate the role of saline on cranial hemodynamic and headache in healthy volunteers.
  Interventions: Drug: Vasoactive Intestinal Peptide (VIP) and Saline

INTERVENTIONS:
Drug: Vasoactive Intestinal Peptide (VIP) and Saline — 12 healthy volunteers of both genders will be included in the main study. Participants will meet twice, with at least one week in between. The main study is a double-blind, randomized, cross-over trial among placebo (sterile saline, non-active substance) and VIP. Intravenous infusion of VIP / placebo (saline) will be conducted over 120 minutes. Patients will be asked after each trial day to record headache strength, accompanying symptoms, and drug use for up to 24 post-infusion.

SUMMARY:
Vasoactive intestinal peptide (VIP) is a peptide of 28 amino acid residues that belongs to the glucagon/secretin superfamily of peptides. It is produced in different regions of the nervous system, including the brain, trigeminovascular system and several autonomic nerves. Once released from neurons, it acts on vasoactive intestinal peptide receptor 1 (VPAC1), vasoactive intestinal peptide receptor 2 (VPAC2) and pituitary adenylate cyclase-activating polypeptide type I receptor (PAC1), by mediating smooth muscle relaxation, vasodilation and water secretion. Along with other neuropeptides, such as calcitonin gene-related peptide (CGRP) and pituitary adenylate cyclase-activating polypeptide (PACAP), it is released from the trigeminal afferents and exerts a strong vasodilating activity on the cranial vasculature, sharing the activation of adenylate cyclase. Especially, it shares 70% structure with PACAP and acts on the same receptors. But, unlike it, VIP cannot induce a long-lasting vasodilation and has a modest capability to induce migraine attacks. Whether a long-lasting infusion of VIP may induce a prolonged vasodilation in the cerebral vessels and migraine, as a twenty-minute infusion of PACAP, is unknown.

ELIGIBILITY:
Inclusion Criteria:

18-60 years. 50-90 kg. Women of childbearing potential must use adequate contraception.

Exclusion Criteria:

Headache less than 48 hours before the tests start All primary headaches Daily consumption of drugs of any kind other than oral contraceptives Pregnant or nursing women. A cardiovascular disease of any kind, including cerebrovascular diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in cranial hemodynamic | Before (-10 minutes) and after infusion (+2 hours) of VIP compared with before and after infusion of saline]
  Change on diameter of superficial temporal artery. Change on diameter will be measured with milletimeter.
Occurrence and change of headache | [Time Frame: Before (-10 minutes) and after infusion (+12 hours) of maxipost compared with before and after infusion of saline]
  Occurrence of headache measured by numerical rating scale (NRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Danish headache center, København S, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pellesi L, Al-Karagholi MA, De Icco R, Chaudhry BA, Lopez CL, Snellman J, Hannibal J, Amin FM, Ashina M. Plasma Levels of CGRP During a 2-h Infusion of VIP in Healthy Volunteers and Patients With Migraine: An Exploratory Study. Front Neurol. 2022 Apr 1;13:871176. doi: 10.3389/fneur.2022.871176. eCollection 2022. PMID 35432170
- [Derived] Pellesi L, Al-Karagholi MA, Chaudhry BA, Lopez CL, Snellman J, Hannibal J, Amin FM, Ashina M. Two-hour infusion of vasoactive intestinal polypeptide induces delayed headache and extracranial vasodilation in healthy volunteers. Cephalalgia. 2020 Oct;40(11):1212-1223. doi: 10.1177/0333102420937655. Epub 2020 Jun 27. PMID 32594760